CLINICAL TRIAL: NCT03092713
Title: The Effect Evaluation of Combined Cognitive and Vocational Interventions After Mild-to-moderate Traumatic Brain Injury: a Randomized Controlled Trial and Qualitative Process Evaluation
Brief Title: Combined Cognitive and Vocational Interventions After Mild-to-moderate TBI: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other); Sunnaas Rehabilitation Hospital (Other); Oslo Metropolitan University (Other); Norwegian Labour and Welfare Administration (Other)
Responsible Party: Principal Investigator, Nada Andelic, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/2038
Record Dates: First submitted 2017-03-10; First posted 2017-03-28 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Brain Injuries, Traumatic; Cognitive Impairment
Keywords: Cognitive Rehabilitation; Supported employment; Mild and moderate TBI; Return to work; Randomized Controlled Trial
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction; Lymphoma, Follicular | interventions — Rehabilitation, Vocational; Employment, Supported; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with active treatment group compared to treatment as usual
Who Masked: Participant, Outcomes Assessor
Masking Description: Particpant are blinded to Group allocation, and all assessments are blinded to Group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Intervention and Supported Employment (CCI-SE) (Active Comparator): Combined cognitive and vocational rehabilitation in a mixed design.
  Interventions: Behavioral: Combined cognitive (Compensatory Cognitive Training - CCT) and vocational rehabilitation (Supported Employment)
- Control group (Active Comparator): Usual follow-up assessment and treatment provided by the multidisciplinary TBI rehabilitation team.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Combined cognitive (Compensatory Cognitive Training - CCT) and vocational rehabilitation (Supported Employment) — The CCI-SE Group receives a manualized Group-based cognitive psycho-educational intervention (10 sessions), combined with supported employment at their work-place.
  Arms: Cognitive Intervention and Supported Employment (CCI-SE)
Behavioral: Control Group — The Control Group receives usual assessment and treatment at Oslo University Hospital.
  Arms: Control group

SUMMARY:
A considerable number of patients with mild and moderate traumatic brain injury (TBI) experience long-lasting somatic, cognitive, and emotional symptoms that may hamper their capacity to return to work (RTW). Although several studies have described medical, psychological and work-related factors that predict RTW after TBI, well-controlled intervention studies regarding RTW in this group are scarce. Furthermore, there have traditionally been weak collaborations among rehabilitation services in the health sector, the Labor and Welfare Administration (NAV), and the work-places.

The current project proposal describes an innovative randomized controlled trial (RCT) which will explore the effect of combined manualized cognitive rehabilitation efforts and supported employment in real-life competitive work settings for patients who have not returned to work 8 weeks post-injury. The project combines the rehabilitation and vocational science perspectives; it involves multidisciplinary collaboration, and explores the efficacy of increased cross-sectorial collaboration between specialized health care services and the welfare system. If the intervention proves efficient, the project will further describe the cost-effectiveness and utility of the program, and thereby provide important information of use for policy makers. In addition, the study aims at generating knowledge on the RTW-process both for the persons with TBI, and their workplaces, and to disseminate this knowledge in order to create new multidisciplinary and collaborative practices. The project has potential to generate knowledge of relevance for other patients with neurological deficit.

DETAILED DESCRIPTION:
Please, see protocol article: https://www.ncbi.nlm.nih.gov/pubmed/29041954

ELIGIBILITY:
Inclusion Criteria:

* reside in Oslo and Akershus counties in Norway
* mild-to-moderate TBI (Glasgow Coma scale score 10-15 at injury site). Confirmation of diagnosis of mild TBI will be done through documenting that acute symptoms adhere to the American Congress of Rehabilitation Medicine's (ACRM) definition of mild TBI.
* loss of consciousness <24 hours
* posttraumatic amnesia (PTA) <7 days
* employed in a minimum 50% position at the time of injury
* sick listed at the 50% or higher level due to post-concussive symptoms 2 months post-injury

Exclusion Criteria:

* history of severe psychiatric or neurological illness
* active substance abuse
* inability to speak and read Norwegian

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Return to work | 18 months post injury
  The effect of the intervention on return to work rates throughout the follow-up period
Work stability | 18 months post injury
  The effect of the intervention on work stability rates throughout the follow-up period

SECONDARY OUTCOMES:
Rivermead post-concussion questionnaire | 18 months
  Questionnaire; The effect of the study intervention on post concussive symptoms
Euro-Qol - 5D (EQ-5D) | 18 months
  Questionnaire; The effect of the study intervention on health-related quality-of-life throughout the follow-up period
Quality of life after brain injury (Qolibri) | 18 months
  Questionnaire; The effect of the study intervention on disease-related quality-of-life throughout the follow-up period

OTHER OUTCOMES:
Fatigue Severity Scale | 18 months
  Questionnaire; The effect of the study intervention on fatigue throughout the follow-up period
Insomnia Severity Index | 18 months
  Questionnaire; The effect of the study intervention on sleep throughout the follow-up period
Cognitive Failures Questionnaire | 18 months
  Questionnaire; The effect of the study intervention on self-reported cogntiive symptoms throughout the follow-up period
Generalized Anxiety Disorder (GAD-7) | 18 months
  Questionnaire; The effect of the study intervention on anxiety throughout the follow-up period
Patient Health Questionnaire (PHQ-9) | 18 months
  Questionnaire; The effect of the study intervention on depression throughout the follow-up period
General Self-efficacy Scale | 18 months
  Questionnaire; The effect of the study intervention on self-efficacy throughout the follow-up period
Neuropsychological functioning | 18 months
  Screening test battery including measures of general ability Level, attention, Processing speed, Learning and memory executive functioning, and performance validity

CONTACTS AND LOCATIONS:
Overall Officials: Nada Andelic, MD; PhD, Principal Investigator — Oslo University Hospital/University of Oslo
Locations (1):
- Oslo University Hospital, Dept. of physical medicine and rehabilitation, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howe EI, Andelic N, Fure SCR, Roe C, Soberg HL, Hellstrom T, Spjelkavik O, Enehaug H, Lu J, Ugelstad H, Lovstad M, Aas E. Cost-effectiveness analysis of combined cognitive and vocational rehabilitation in patients with mild-to-moderate TBI: results from a randomized controlled trial. BMC Health Serv Res. 2022 Feb 12;22(1):185. doi: 10.1186/s12913-022-07585-3. PMID 35151285
- [Derived] Howe EI, Fure SCR, Lovstad M, Enehaug H, Sagstad K, Hellstrom T, Brunborg C, Roe C, Nordenmark TH, Soberg HL, Twamley E, Lu J, Andelic N. Effectiveness of Combining Compensatory Cognitive Training and Vocational Intervention vs. Treatment as Usual on Return to Work Following Mild-to-Moderate Traumatic Brain Injury: Interim Analysis at 3 and 6 Month Follow-Up. Front Neurol. 2020 Nov 10;11:561400. doi: 10.3389/fneur.2020.561400. eCollection 2020. PMID 33240196
- [Derived] Howe EI, Langlo KS, Terjesen HCA, Roe C, Schanke AK, Soberg HL, Sveen U, Aas E, Enehaug H, Alves DE, Klethagen P, Sagstad K, Moen CM, Torsteinsbrend K, Linnestad AM, Nordenmark TH, Rismyhr BS, Wangen G, Lu J, Ponsford J, Twamley EW, Ugelstad H, Spjelkavik O, Lovstad M, Andelic N. Combined cognitive and vocational interventions after mild to moderate traumatic brain injury: study protocol for a randomized controlled trial. Trials. 2017 Oct 17;18(1):483. doi: 10.1186/s13063-017-2218-7. PMID 29041954
- See also: Protocol paper — https://www.ncbi.nlm.nih.gov/pubmed/29041954
- See also: Baseline paper — http://pubmed.ncbi.nlm.nih.gov/34314269/
- See also: The interim analysis paper — http://pubmed.ncbi.nlm.nih.gov/33240196/
- See also: The intervention effect paper — http://pubmed.ncbi.nlm.nih.gov/33957293/